CLINICAL TRIAL: NCT06858501
Title: Concordance in Response Assessment Incorporating Meta-Iodobenzylguanidine (123I-MIBG) and Meta-[18F]Fluorobenzylguanidine (18F-MFBG, IND#146379, NSC#853868) Imaging in Neuroblastoma
Brief Title: Comparing 123I-MIBG and 18F-MFBG Imaging in Patients With Newly Diagnosed, High Risk Neuroblastoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PEPN24N1; NCI-2025-00042 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEPN24N1 (Other: Pediatric Early Phase Clinical Trial Network); PEPN24N1 (Other: CTEP); UM1CA228823 (NIH)
Record Dates: First submitted 2025-01-23; First posted 2025-03-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Ganglioneuroblastoma; Ganglioneuroblastoma, Nodular; High Risk Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma | interventions — Specimen Handling; 3-fluorobenzylguanidine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Diagnostic (18F-MFBG) (Experimental): Patients receive 18F-MFBG IV over 1 minute and undergo PET/CT or PET/MRI over 9-30 minutes at the time of each SOC 123I-MIBG scan (at the time of induction cycle 1, at the end of the last induction cycle, and at the time of first relapse/disease progression).
  Patients may undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Florbenguane F18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Florbenguane F18 — Given IV
  Other Names: 18F meta-Fluoro Benzylguanidine; 18F-MFBG; [(18)F]-MFBG; Florbenguane (18F); FLORBENGUANE F-18; IRP 101; IRP-101; meta-[(18)F]-Fluorobenzylguanidine; meta-Fluorine F 18 Fluorobenzylguanidine; Meta-fluoro Benzylguanidine F-18
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT or PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial evaluates whether an investigational scan (18F-MFBG positron emission tomography [PET]/computed tomography [CT] or PET/magnetic resonance imaging [MRI]) can accurately detect tumors in patients with newly diagnosed, high-risk neuroblastoma as well as standard of care imaging with 123 I-MIBG. 18F-MFBG is a radioactive diagnostic agent that is injected into a vein and taken up by tumor cells. The cells can then be visualized using PET/CT or PET/MRI scans. A PET scan uses radioactive material injected into the blood to show the internal workings of the body. A CT scan uses x-rays and a computer to produce a 3-dimensional image of the body. MRI uses radiofrequency waves and a strong magnetic field rather than x-rays to provide clear and detailed pictures of internal organs and tissues. Combining PET with CT or MRI may help doctors better understand the extent and the exact location of disease. Diagnostic procedures, such as 18F-MFBG PET/CT or PET/MRI, may detect tumors as well as or better than the current standard imaging with 123 I-MIBG in patients with newly diagnosed, high-risk neuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the concordance in International Neuroblastoma Response Criteria (INRC) response designations at the end of induction as assessed by iobenguane I-123 (123I-MIBG) and florbenguane F18 (18F-MFBG) central reads in patients with high-risk stage L2 and stage M neuroblastoma.

SECONDARY OBJECTIVES:

I. To describe individual metastatic lesion response using 123I-MIBG and 18F-MFBG imaging at diagnosis and end-induction.

II. To describe concordance in central Curie score between 123I-MIBG and 18F-MFBG imaging.

III. To describe concordance in end of induction response designations (poor end-of induction response versus [vs.] good end-of induction response) as assessed by 123I-MIBG and 18F-MFBG in patients receiving high-risk therapy.

IV. To describe concordance as assessed by 123I-MIBG and 18F-MFBG in the INRC components of primary (soft tissue) tumor response and tumor response at metastatic soft tissue and bone sites in patients receiving high-risk therapy.

EXPLORATORY OBJECTIVES:

I. To describe concordance in International Neuroblastoma Risk Group Staging System (INRGSS) stage as assessed by 123I-MIBG and 18F-MFBG.

II. To describe the natural history of discordant lesions detected only by 18F-MFBG and not by 123I-MIBG in patients with high-risk neuroblastoma, and to describe additional interventions undertaken (including additional imaging, biopsies, and/or additional therapies) based on identification of discordant lesions.

III. To describe the change in standardized uptake value (SUV) of the primary and metastatic lesions on 18F-MFBG scans from diagnosis to end of induction.

IV. To evaluate the patient/family experience with 123I-MIBG and 18F-MFBG imaging.

V. To describe concordance between detection of disease using 123I-MIBG imaging (Curie score), 18F-MFBG imaging (Curie score) and the percentage of circulating tumor deoxyribonucleic acid (DNA) (as a continuous variable) testing during high-risk neuroblastoma therapy.

VI. To identify logistical barriers to successful imaging using 18F-MFBG. VII. To quantify inter-observer variability of Curie scores on 18F-MFBG and 123I-MIBG among central reviewers.

VIII. To describe acute toxicity of 18F-MFBG administration. IX. To estimate the progression free survival (PFS) and overall survival (OS) among eligible patients enrolled on the study.

OUTLINE:

Patients receive 18F-MFBG intravenously (IV) over 1 minute and undergo PET/CT or PET/MRI over 9-30 minutes at the time of each standard of care (SOC) 123I-MIBG scan (at the time of induction cycle 1, at the end of the last induction cycle, and at the time of first relapse/disease progression). Patients may undergo blood sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Any age at diagnosis.
* Patients must have a diagnosis of neuroblastoma or ganglioneuroblastoma (nodular, unfavorable subtype) verified by tumor pathology analysis or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites.
* Patients must have high-risk neuroblastoma defined as one of the following:

  * Any age with International Neuroblastoma Risk Group (INRG) stage L2 or M and MYCN amplification.
  * Age ≥ 547 days and INRG stage M regardless of biologic features.
  * Age ≥ 547 days and INRG stage L2 with unfavorable histology.
* Patients must have newly diagnosed disease.
* Patients must have either measurable or evaluable disease by INRC.
* Patients observed or treated with a single cycle of chemotherapy per a low- or intermediate-risk neuroblastoma regimen (e.g. as per ANBL0531, ANBL1232 or similar) for what initially appeared to be non-high-risk disease, but subsequently found to meet high-risk criteria will be eligible. These patients must enroll prior to the start of high-risk therapy.
* Patients who receive localized emergency radiation to sites of life-threatening or function-threatening disease prior to or immediately after establishment of the definitive diagnosis will be eligible.
* Patients initially recognized to have high-risk disease must enroll prior to or within the first week after starting high-risk induction chemotherapy.
* Induction therapy as per a standard high-risk neuroblastoma induction regimen (examples include ANBL1531 arm A, ANBL2131 arm A, or ANBL2131 arm B) must be planned for patients to be eligible for this study.

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events of radiation. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control, including a medically accepted barrier or contraceptive method (e.g., male or female condom) at least 48 hours prior to and following all imaging studies. Abstinence is an acceptable method of birth control.
* Norepinephrine transporter (NET)-dependent agents: Many medications are known to interfere with uptake of NET-dependent agents. Investigators should use caution when prescribing these medications for patients undergoing procedures on this study. Medications that are known to substantially interfere with uptake of NET-dependent agents should be held if possible, based on patient condition 24 hours prior to each 18F-MFBG scan. These agents can be resumed immediately after each 18F-MFBG scan is completed. Patients who are receiving medications that are known to significantly interfere with uptake of NET-dependent agents (primarily tricyclic antidepressants, psychostimulants, and antihypertensives) and for whom these medications cannot be safely withheld before the start of study procedures will not be eligible.
* The patient has a known or suspected history of significant allergic reaction or anaphylaxis to any components of the 18F-MFBG or 123I-MIBG imaging agents.
* Patients who will require sedation or anesthesia only for 18F-MFBG imaging.

  * Note: Patients who need anesthesia will be required to have 18F-MFBG imaging combined with other scans or procedures necessary for clinical care (ex: MRI, bone marrow aspirate/biopsies, line placement).
* Patients will be able to enroll prior to baseline 123I-MIBG imaging. However, patients who have had their baseline standard of care 123I-MIBG imaging prior to enrollment who have known MIBG non-avid disease are not eligible.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-03-22 (Estimated); Primary Completion 2028-12-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Concordance in International Neuroblastoma Response Criteria (INRC) objective response measures | Up to 105 days
  Will be estimated with 95% confidence intervals (CIs) using the unweighted kappa coefficient at each of the three time points.

SECONDARY OUTCOMES:
Individual metastatic lesion response | Up to 105 days
  Will be assessed using iobenguane I-123 (123I-MIBG) and florbenguane F18 (18F-MFBG) imaging. Response will be summarized by number (percent [%]) of lesions stratified by imaging modality. A generalized linear mixed model will also estimate percent response by imaging modalities and compare response between modalities. The model will include fixed effects for modality, cumulative logit link function, multinomial distribution, and random effects for patient and lesion within patient.
Curie scores | Up to 3 years
  Will estimate the correlation between Curie scores on both 123I-MIBG and 18F-MFBG imaging using Spearman rank correlation with a 95% CI.
Concordance in end of induction response | Up to 105 days
  Will be measured as poor versus good. Will be assessed by 123I-MIBG and 18F-MFBG in patients receiving high-risk therapy. Will be estimated by the kappa coefficient.
Concordance in 123I-MIBG and 18F-MFBG scans by INRC components | Up to 105 days
  Will be assessed by primary (soft tissue) tumor response and tumor response at metastatic soft tissue and bone sites, in patients receiving high-risk therapy. Concordance will be estimated using Cohen's kappa.

OTHER OUTCOMES:
Concordance in International Neuroblastoma Risk Group Staging System (INRGSS) stage | Up to 3 years
  Will be assessed by 123I-MIBG and 18F-MFBG. Will be estimated by the unweighted kappa coefficient and Cicchetti-Allison weight kappa coefficient with 95% confidence intervals.
Natural history of discordant lesions | Up to 3 years
  Will be assessed only by 18F-MFBG and not by 123I-MIBG in patients with high-risk neuroblastoma. The natural history of disease sites detected by 18F-MFBG and 123I-MIBG at diagnosis and during therapy will be evaluated in a patterns of failure analysis. Specific disease sites detected at relapse will be coded as having been identified by 18F-MFBG, 123I-MIBG, neither scan or both scans at diagnosis and at end of induction. The number of individual sites identified at relapse that were detected previously by 18F-MFBG, 123I-MIBG, neither or both scans will be tabulated and the proportion of sites detected by each scan type will be reported.
Additional interventions undertaken based on identification of discordant lesions | Up to 3 years
  Frequency of additional interventions undertaken based on identification of discordant lesions including additional imaging, biopsies, and additional therapies.
Change in standardized uptake value (SUV) of the primary and metastatic lesions | Up to 105 days
  Will be estimated using a general linear mixed model. The model will include fixed effects for lesion type (primary/metastatic), imaging modality, and the lesion type-imaging interaction term. The model will also include random effects for patient and lesion within patient. Contrasts will be specified to estimate the mean change in SUV between primary and metastatic lesions by imaging modality.
Patient/family experience with 123I-MIBG and 18F-MFBG imaging | Up to 3 years
  An optional study that will be completed using the Patient Family Questionnaire. Will assess survey answers based on the symptoms and experiences that occur within 24 hours of the scan.
Percentage of circulating tumor deoxyribonucleic acid (DNA) | Up to 3 years
  Spearman rank correlation will estimate the correlation between the Curie scores and percentage of circulating tumor DNA stratified by imaging modality.
Logistical barriers to successful imaging using 18F-MFBG | Up to 3 years
  Will be assessed using descriptive summary. The reasons for incomplete imaging, per protocol, will be collected in the study case report forms and summarized by frequencies with percentages.
Inter-observer variability of Curie scores | Up to 3 years
  Intraclass correlation coefficients (ICC) will estimate proportion of variances in Curie scores attributable to central reviewers. A general linear mixed model with random effects for patient, reviewer, and patient-reviewer interaction will estimate the ICC.
Incidence of acute toxicity of 18F-MFBG administration | Up to 3 years
  Acute toxicities will be summarized by frequencies with percentages.
Progression free survival | Up to 3 years
  Kaplan-Meier curves will estimate median (95% CI) time to progression.
Overall survival | Up to 3 years
  Kaplan-Meier curves will estimate median (95% CI) time to death.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya C Watt, Principal Investigator — Pediatric Early Phase Clinical Trial Network